CLINICAL TRIAL: NCT06504420
Title: A Randomized, Multicenter, Double-blind, Placeobo-control Study of Sirolimus for Primary Antiphospholipid Syndrome Patients
Brief Title: The Safety and Efficiency of Sirolimus in Primary Antiphospholipid Syndrome: a Randomized Control Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Zhanguo Li, Department of Rheumatology and immunology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20240125
Record Dates: First submitted 2024-07-11; First posted 2024-07-16 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Primary Antiphospholipid Syndrome
Keywords: APS
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sirolimus (Experimental): Sirolimus 1.5mg po. QD
  Interventions: Drug: Sirolimus
- placeobo (Placebo Comparator): Sirolimus placebo 1.5mg po. QD
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sirolimus — Subjects will receive Sirolimus 1.5mg/d for 48 weeks in addition to their ongoing APS treatment regimen
  Arms: Sirolimus
Drug: Placebo — Subjects will receive Placebo 1.5mg/d for first 24 weeks and Sirolimus 1.5mg/d for next 24 weeks in addition to their ongoing APS treatment regimen
  Arms: placeobo

SUMMARY:
This study is an Investigator initiated, randomized, multicenter, double-blind, placebo-control study. The aim of this study is to evaluate the safety and efficiency of Sirolimus for primaty antiphospholipid syndrome patients at week 24 and week 48.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and sign the informed consent form
2. Male or Female
3. aged 18-70 at the time of screening visit
4. Met 2006 Sapporo classification criteria of APS or 2023 ACR/EULAR classification criteria of APS
5. With the stable combination therapy

Exclusion Criteria:

1. history of serious adverse events or contraindication to Sirolimus
2. Catastrophic APS within 90 days
3. Acute thrombosis within 30 days
4. ≥4/11 American College of Rheumatology Classification Criteria for SLE or other systemic autoimmune diseases
5. Historically positive HIV test or test positive at screening for HIV
6. currently on any suppressive therapy for a chronic infection (such as tuberculosis, hepatitis B infection, hepatitis C infection, CMV, EBV, Syphilis, etc)
7. Surgery treatment within one month
8. History of malignant neoplasm within the last 5 years
9. White blood cell counts<3×10*9/L
10. Abnormal Liver function tests: ALT or AST ≥ 1.5 times the upper limit of the normal value, and total bilirubin and blood lipids ≥ 2 times the upper limit of the normal value
11. Pregnant or pregnancy preparation or breastfeed
12. Any circumstances that may cause the subjects to be unable to complete the study or pose significant risks to the subjects

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Complete response(CR) rate at week 24 | week 24
  CR will be defined as follows: 1.No thrombosis events; 2.PLT ≥100 and with nobleeding; 3. No persistent autoimmnune haemolytic anaemia; 4. No skin ulcer; 5.No renal thrombotic microangiopathy; 5.Normal cognitive function (MoCA score ≥26）.
Partial response (PR) rate at week 24 | week 24
  PR will be defined as one of follows: 1.superficial thrombotic events;2. PLT ≥30 or increased at least 2 times of baseline and with no bleeding;3.haemoglobulin concentration normal or increased 20g/L compared to baseline; 4.50% improvement; 5. a serum creatinine level 15% abov baseline, RBCs per high-power field 50% above baseline with no casts, 50% improvement in the urinary prt:cr; 6. milde cognitive diysfunction (MoCA 9~25).

SECONDARY OUTCOMES:
Complete response(CR) rate at week 48 | week 48
  CR will be defined as follows: 1.No thrombosis events; 2.PLT ≥100 and with nobleeding; 3. No persistent autoimmnune haemolytic anaemia; 4. No skin ulcer; 5.No renal thrombotic microangiopathy; 5.Normal cognitive function (MoCA score ≥26）.
Partial response (PR) rate at week 48 | week 48
  PR will be defined as one of follows: 1.superficial thrombotic events;2. PLT ≥30 or increased at least 2 times of baseline and with no bleeding;3.haemoglobulin concentration normal or increased 20g/L compared to baseline; 4.50% improvement; 5. a serum creatinine level 15% abov baseline, RBCs per high-power field 50% above baseline with no casts, 50% improvement in the urinary prt:cr; 6. milde cognitive diysfunction (MoCA 9~25).
Rate of Participants with adverse effects and serious adverse effects during treatment | baseline to week 48
  Adverse effects include fever, rash, abnormal liver function, rate of new-onset infections and any abnormal measures after recivede study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, Study Director — Peking university peoples hospital

IPD SHARING:
Plan to Share IPD: No